CLINICAL TRIAL: NCT01244854
Title: Life Goals Behavioral Change to Improve Outcomes for Veterans With SMI
Brief Title: Life Goals Behavioral Change to Improve Outcomes for Veterans With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RRP 10-226
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Bipolar Disorder; Schizophrenia; Major Depressive Disorder; Chronic Affective Disorders; Cardiovascular Disease Risk
Keywords: chronic mental disorders; cardiovascular disease; behavior change
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Depressive Disorder, Major; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): Enhanced Usual Care; patients receive care as usual, with additional mailings on wellness newsletter topics
  Interventions: Behavioral: Life Goals Collaborative Care

INTERVENTIONS:
Behavioral: Life Goals Collaborative Care — LGCC consists of 1) 10 sessions focused on CVD risk reduction through behavioral change within the context of patients' psychiatric symptoms; 2) participant goal setting in diet and exercise; 3) customized ongoing motivational interviewing (MI)-based patient contacts with a health specialist for 6 months, in addition to 4) strategies to increase provider access and support for behavioral change and medical management.

SUMMARY:
Persons with serious mental illness are at increased risk of cardiovascular disease. The goals of this study are to test a treatment, Life Goals Collaborative Care to help promote health behavior change and to get feedback from patients and providers on what is needed to help better coordinate and physical and mental health care of these patients.

DETAILED DESCRIPTION:
Background: Persons with serious mental illness (SMI, including schizophrenia, bipolar disorder, or chronic affective disorders) experience a disproportionate burden of medical comorbidity, notably cardiovascular disease (CVD), leading to poor functioning and premature mortality. CVD risk factors in persons with SMI are attributable to unhealthy lifestyles exacerbated by mental health-related symptoms, medication side effects (e.g., weight gain), and the fragmentation of physical and mental health services.

Objectives: The specific aims of this rapid response proposal pilot study are 1) to adopt and test the feasibility of an evidence-based psychosocial intervention (Life Goals Collaborative Care- or LGCC) designed to promote health behavioral change that was developed for bipolar disorder to a broader SMI patient population, and 2) to describe the implementation of LGCC and the barriers and facilitators of adoption to a more generalizable SMI patient population, and to vet the program to key VA stakeholders in order to inform a larger implementation study across different VHA settings.

Methods: LGCC is a novel manual-based intervention that incorporates behavioral change strategies within a Chronic Care Model-based program. It is designed to reduce risk factors for cardiovascular disease (CVD), through improved control of psychiatric symptoms and increased positive health behaviors, as well as improved coordination of physical and mental health care. We will enroll 100 individuals diagnosed with a chronic mental disorder and CVD risk factor who are also receiving care within the VA Ann Arbor Healthcare System mental health clinics, of which 50 will be randomized to LGCC, and 50 randomized to receive usual care. LGCC consists of 1) 10 sessions focused on CVD risk reduction through behavioral change within the context of patients' psychiatric symptoms; 2) participant goal setting in diet and exercise; 3) customized ongoing motivational interviewing (MI)-based patient contacts with a health specialist for 6 months, in addition to 4) strategies to increase provider access and support for behavioral change and medical management. Outcomes will be assessed to determine whether effect sizes are comparable to previously published LGCC randomized controlled trials, and include mental and physical health-related quality of life and long-term (10-year) CVD risk based on the Framingham risk score assessed at 6 months. Additional mixed methods analyses of administrator, consumer and provider interviews to inform further adoption of LGCC will also be completed.

Impact: Serious mental illness is associated with significant disability, decreased quality of life, and a decreased life span. VA patients with SMI die an average of 13-18 years earlier than age and gender matched individuals from the U.S. population, mostly from CVD. Interventions such as LGCC that combine individualized lifestyle coaching with Chronic Care Model principles may lead to the greatest impact on this public health crisis because they address multiple reasons for health disparities, and behavior change is reinforced through improved coordination and continuity of care. If effective, LGCC could be easily disseminated in VA practices and aligned with emerging VHA "T-21" initiatives around veteran-centered care (patient-centered medical home) and behavioral medicine programs that can ultimately improve outcomes for veterans with mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of serious mental illness (schizophrenia, bipolar disorder, other psychosis, major depressive disorder, or other recurrent depression or affective disorder)
* Have at least one of the following risk factors for CVD (cardiovascular disease):

Body mass index (BMI) >28 or waist circumference of >35 (women) or >40 (men) inches OR Self-reported diagnosis of hypertension ("high blood pressure"), dyslipidemia ("high cholesterol") or diabetes or high blood sugar OR Documentation in the medical record of a diagnosis of or treatment for hypertension (defined as documented diagnosis or blood pressure of >140/90 on 2 occasions or prescription for an antihypertensive medication), dyslipidemia (documented diagnosis or LDL>160 or prescription for a lipid-lowering medication) or diabetes mellitus (documented diagnosis or HbA1C >7% or current prescription for oral hypoglycemic therapy)

Exclusion Criteria:

* Have unresolved substance intoxication or withdrawal, such as appearing to be intoxicated (e.g., incoherent, slurred speech), or experiencing withdrawal symptoms from substance abuse at the time of enrollment.
* Are unwilling or unable to provide informed consent or comply with study requirements at the time of enrollment (e.g., unable to complete forms or attend sessions due to substantial functional limitations).
* Active suicidal ideation at time of enrollment (focused interventions are more appropriate for this group)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2012-08-13 (Actual); Study Completion 2015-03-06 (Actual)

PRIMARY OUTCOMES:
overall health-related quality of life | 6 months

SECONDARY OUTCOMES:
Framingham risk score | 6 months
total cholesterol | 6 months
systolic blood pressure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy M. Kilbourne, PhD MPH, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Goodrich DE, Lai Z, Lasky E, Burghardt AR, Kilbourne AM. Access to weight loss counseling services among patients with bipolar disorder. J Affect Disord. 2010 Oct;126(1-2):75-9. doi: 10.1016/j.jad.2010.02.138. Epub 2010 Apr 8. PMID 20381155
- [Result] Kilbourne AM, Bramlet M, Barbaresso MM, Nord KM, Goodrich DE, Lai Z, Post EP, Almirall D, Verchinina L, Duffy SA, Bauer MS. SMI life goals: description of a randomized trial of a collaborative care model to improve outcomes for persons with serious mental illness. Contemp Clin Trials. 2014 Sep;39(1):74-85. doi: 10.1016/j.cct.2014.07.007. Epub 2014 Jul 30. PMID 25083802
- [Derived] Kilbourne AM, Barbaresso MM, Lai Z, Nord KM, Bramlet M, Goodrich DE, Post EP, Almirall D, Bauer MS. Improving Physical Health in Patients With Chronic Mental Disorders: Twelve-Month Results From a Randomized Controlled Collaborative Care Trial. J Clin Psychiatry. 2017 Jan;78(1):129-137. doi: 10.4088/JCP.15m10301. PMID 27780336